CLINICAL TRIAL: NCT03600285
Title: Prospective, Single-Arm, Study to Assess the Safety and Performance of the TB1-K Device for Organ Preservation in Donor Kidneys for Transplantation
Acronym: EMERGE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Transplant Biomedicals, S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TB/TB1K-001
Record Dates: First submitted 2018-07-06; First posted 2018-07-26 (Actual); Last update posted 2019-06-21 (Actual); Status verified 2019-06

CONDITIONS: Kidney Preservation and Transportation
Keywords: VIVIAN

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TB1-K (Experimental): TB1-K preservation arm
  Interventions: Device: TB1-K

INTERVENTIONS:
Device: TB1-K — Use of TB1-K for preservation and transport of donated kidneys

SUMMARY:
TB1-K Device is an organ preservation and transportation system, using ultrasound technology with a cooling system to preserve the organ in optimal conditions during transport to the transplant recipient.

This is a prospective, single-arm, multi-center study comparing to a historical control for cold storage.

The study is conducted in accordance with the Standard ISO 14155 (Clinical investigation of medical devices for human subjects - Good clinical practice), and other legal requirements.

The study objective is to assess the safety and performance of the TB1-K device in donor kidneys intended for transplantation.

ELIGIBILITY:
Donor Inclusion Criteria:

1. Donor kidney suitable for preservation
2. Only one kidney per donor will be included
3. Cold ischemia time (CIT) ≤ 24 hours
4. Donor age over 18 years old
5. Donor meets one of the following:

   1. Donor after brain death (DBD), standard and extended criteria
   2. Donor after circulatory death (DCD), cardiac arrest Maastricht classification III (awaiting cardiac arrest, controlled)
6. Signed written informed consent

Donor Exclusion Criteria:

1. Kidney, which investigator is unwilling to use, or presence of moderate or severe traumatic kidney injury, or anatomical kidney vascular abnormalities, which would preclude the organ from being acceptable by the transplant surgeon
2. Donor after circulatory death (DCD), Maastricht classification I, II, IV, V (See Definitions, section 14)
3. Living donors
4. Previous usage of a perfusion machine (PM)
5. Kidneys not considered suitable for preservations
6. Positive serology (HIV, Hepatitis B surface antigen & C)

Recipient Inclusion Criteria:

1. Registered primary kidney transplant candidate, male or female
2. Age ≥ 18 years old
3. Signed written informed consent

Recipient Exclusion Criteria:

1. Prior solid organ or bone marrow transplant
2. Multi-organ transplant
3. Active malignancy
4. Active infection
5. Pregnant females, females intending to get pregnant, or not willing to use a secure contraceptive method.
6. Participation in another clinical trial.
7. Patient with known donor-specific HLA antibody

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-06-29 (Actual); Primary Completion 2019-02-15 (Actual); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
Rate of DGF | 1 week after transplant
  Rate of delayed graft function (DGF), defined as need for dialysis in the first week after transplant, once hyperacute rejection, vascular and urinary tract complications are ruled out.

CONTACTS AND LOCATIONS:
Overall Officials: Fritz Diekmann, PhD, Principal Investigator — Hospital Clinic i provincial de Barcelona
Locations (3):
- Spain (3):
  - Hospital Unviersitario de Bellvitge, Barcelona, Hospitalet de Llobregat
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Clinic i Provincial de Barcelona, Barcelona

IPD SHARING:
Plan to Share IPD: No